CLINICAL TRIAL: NCT00688779
Title: A Double Blind, Placebo Controlled, Randomised, First Time In Man. Study to Investigate the Tolerability, Safety, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of AZD8848 Administered Intranasally to Healthy Male Volunteers and Seasonal Allergic Rhinitis Male Patients Out Of Season
Brief Title: Tolerability/Safety of Intranasal AZD8848 in Healthy Male Volunteers and Seasonal Allergic Rhinitis Male Patients Out of Season
Acronym: SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0540C00001
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Healthy; Allergic Rhinitis
Keywords: Healthy male; allergic rhinitis; tolerability; safety; intranasally; Healthy subjects
MeSH Terms: conditions — Rhinitis, Allergic | interventions — AZD8848

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8848
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8848 — Concentrate for nasal spray,solution 60 mg/g
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Investigate safety/tolerability after a single dose intranasal administration of AZD8848 comparator placebo to healthy male volunteers and seasonal allergic rhinitis male patients out of season

ELIGIBILITY:
Inclusion Criteria:

* History of birch and/or timothy grass pollen induced seasonal allergic rhinitis for at least the previous 2 years
* Body mass index (BMI) between 19 and 30 kg/ m2 and a weight between 50 and 100 kg
* No clinically relevant abnormal findings

Exclusion Criteria:

* Acute illness which requires medical intervention
* Definite or suspected personal history of adverse drug reactions or drug hypersensitivity
* Clinical relevant disease or disorder (past or present)
* A history of asthma

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Incidence/nature of adverse events, 12-lead ECG, pulse, BP, body temperature, spirometry | During the study

SECONDARY OUTCOMES:
Clinical chemistry, haematology, urinalysis | During the study
Nasal symptoms and peak nasal inspiratory flow | During the study
Pharmacokinetics | During the study
Biomarkers nasal lavage and blood | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Edward Högestätt, Principal Investigator — Department of Clinical Chemistry and Pharmacology, Department of Laboratory Medicine on University Hospital Lund, Sweden; Leif T Eriksson, Study Director — AstraZeneca R&D, Lund
Locations (1):
- Research Site, Lund, Sweden

REFERENCES:
- [Derived] Greiff L, Cervin A, Ahlstrom-Emanuelsson C, Almqvist G, Andersson M, Dolata J, Eriksson L, Hogestatt E, Kallen A, Norlen P, Sjolin IL, Widegren H. Repeated intranasal TLR7 stimulation reduces allergen responsiveness in allergic rhinitis. Respir Res. 2012 Jun 22;13(1):53. doi: 10.1186/1465-9921-13-53. PMID 22726593
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1656&filename=D0540C00001_Study_Synopsis.pdf